CLINICAL TRIAL: NCT02576301
Title: Ph 1b Dose Escalation Study of OXi4503 as a Single Agent and in Combination With Cytarabine With Subsequent Phase 2 Cohorts for Subjects With Relapsed/Refractory Acute AML and MDS
Brief Title: Dose Escalation of OXi4503 as Single Agent and Combination With Cytarabine w/Subsequent Ph 2 Cohorts for AML and MDS
Acronym: AML
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mateon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OX1222
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2017-09

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndromes
Keywords: AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 2 AML (Experimental): OXi4503 at MTD plus cytarabine 1g/m2/day
  Interventions: Drug: Phase 2 - OXi4503 + cytarabine
- Phase 2 MDS (Experimental): OXi4503 at MTD plus cytarabine 1g/m2/day
  Interventions: Drug: Phase 2 - OXi4503 + cytarabine
- OXi4503 dose escalation (Experimental): MTD for OXi4503 will be determined
  Interventions: Drug: Phase 1 - OXi4503
- OXi4503 + cytarabine dose escalation (Experimental): MTD of the combination of OXi4503 + cytarbine will be determined
  Interventions: Drug: Phase 1 - OXi4503 + cytarabine

INTERVENTIONS:
Drug: Phase 1 - OXi4503 — Determination of MTD of OXi4503
  Other Names: CA1P; combretastatin A1-diphosphate
  Arms: OXi4503 dose escalation
Drug: Phase 1 - OXi4503 + cytarabine — Determination of MTD of the combination of OXi4503 + cytarabine
  Other Names: CA1P; combretastatin A1-diphosphate
  Arms: OXi4503 + cytarabine dose escalation
Drug: Phase 2 - OXi4503 + cytarabine — Safety and efficacy of the combination of OXi4503 + cytarabine in subjects with AML
  Other Names: CA1P; combretastatin A1-diphosphate
  Arms: Phase 2 AML
Drug: Phase 2 - OXi4503 + cytarabine — Safety and efficacy of the combination of OXi4503 + cytarabine in subjects with MDS
  Other Names: CA1P; combretastatin A1-diphosphate
  Arms: Phase 2 MDS

SUMMARY:
Phase 1 will investigate maximum tolerated dose of OXi4503 as a single agent and in combination with intermediate-dose cytarabine in subjects with relapsed/refractory AML or MDS.

Phase 2 will investigate overall response rate of OXi4503 in combination with intermediate-dose cytarabine in 1) subjects with MDS after failure of 1 prior hypomethylating agent (Arm A) and 2) subjects with relapsed and refractory AML after treatment failure of up to 1 prior chemotherapy regimen (Arm B).

DETAILED DESCRIPTION:
Phase 1 dose escalation component will assess the safety, PK/PD, and preliminary efficacy of OXi4503 as a single agent in subjects with relapsed/refractory AML and MDS, and the safety and PK/PD of the combination of OXi4503 with intermediate-dose cytarabine in subjects with AML/MDS.

Phase 2 will assess the preliminary efficacy of the OXi4503+cytarabine combination in 2 cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent
2. ≥ 18 years of age
3. Phase 1 (dose escalation) subjects must have either:

   * AML that has failed to achieve complete remission or morphologic complete remission or
   * MDS - Marrow blasts must be > 5% and disease failed at least 1 prior hypomethylating agent
4. Phase 2 (expansion) subjects must have either MDS or relapsed/refractory AML
5. Eastern Cooperative Oncology Group performance status 0, 1, or 2
6. Total bilirubin ≤ 2
7. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times upper limit of normal (ULN)
8. Serum creatinine < 2.5 times ULN
9. Prothrombin time (PT)/international normalized ratio and (PTT) in normal range ± 25%
10. Women of child-bearing potential
11. Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods

Exclusion Criteria:

1. Acute promyelocytic leukemia
2. Absolute peripheral blood myeloblast count greater than 20,000/mm3
3. Uncontrolled hypertension
4. History of congenital long QT syndrome or torsades de pointes
5. Pathologic bradycardia or heart block
6. Prolonged baseline QTc
7. Hiistory of ventricular arrhythmia
8. Myocardial infarction and/or new ST elevation
9. Any history of hemorrhagic stroke
10. Symptomatic congestive heart failure
11. Major hemorrhagic event within 28 days
12. Suggestive central nervous system involvement with leukemia
13. Any open wound
14. Pregnant and nursing subjects are excluded
15. Treatment with any anticancer therapy
16. Treatment with colchicine is excluded.
17. Psychiatric disorders that would interfere with consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Phase 1b:MTD of OXi4503 as a single agent and in combination with intermediate-dose cytarabine in subjects with relapsed/refractory AML or MDS | 1 year
Phase 2: Overall response rate of OXi4503 in combination with intermediate-dose cytarabine in subjects with MDS after failure of 1 prior hypomethylating agent (Arm A), and subjects with relapsed and refractory AML after treatment failure of up | 2 years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Johnson SP, Ogunlade O, Lythgoe MF, Beard P, Pedley RB. Longitudinal Photoacoustic Imaging of the Pharmacodynamic Effect of Vascular Targeted Therapy on Tumors. Clin Cancer Res. 2019 Dec 15;25(24):7436-7447. doi: 10.1158/1078-0432.CCR-19-0360. Epub 2019 Sep 24. PMID 31551349